CLINICAL TRIAL: NCT02389101
Title: Molecular and Whole-body MR Imaging in Lymphomas
Acronym: MILY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Heikki Minn, Professor, Chief Physician, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T164/2014
Record Dates: First submitted 2014-10-22; First posted 2015-03-17 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin
Keywords: Lymphoma; 68Ga-DOTANOC PET/CT; Somatostatin receptor; MRI; Diffusion weighted imaging; Early treatment response
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lymphoma (Experimental): Newly diagnosed lymphoma, all subtypes allowed
  Interventions: Other: 68Ga-DOTANOC PET/CT; Diffusion weighted MRI

INTERVENTIONS:
Other: 68Ga-DOTANOC PET/CT; Diffusion weighted MRI — PET/CT: Radionuclide imaging using short-lived isotope Ga-68; MRI imaging w/o gadolinium contrast

SUMMARY:
Lymphomas are classified as Hodgkin's or non-Hodgkin's lymphomas, of which especially the latter represent a heterogeneous group with varying patterns of prognosis, biological behaviour and response to treatment. 18F-FDG PET/CT is useful for staging and response monitoring but has the disadvantage of associated radiation exposure which may not be desirable for young patients. Advanced MRI techniques including diffusion weighted imaging (DWI) are increasingly used for improved lesion detection and characterisation of lymphomas and in the whole-body mode offer a promising radiation-free alternative to CT. Molecular imaging in turn is important in theranostics medicine where detection of therapeutic target is essential. The concept of theranostics has been successfully adapted to management of neuroendocrine tumors (NET) where peptide receptor radiotherapy (PRRT) is offered to patients progressing on treatment with long-acting somatostatin analogues.

Recently in the investigator's hospital a case of diffuse large B-cell lymphoma (DLBCL) was initially misdiagnosed as NET because of high uptake of 68Ga-DOTANOC in pancreatic tumor at PET/CT. A PubMed search revealed a similar case report in bronchial tumor which turned out to be DLBCL (Jain et al. Clin Nucl Med 2014;39:358-359). Bearing these two cases in mind the investigators now aim to systematically study somatostatin receptor status (ssr) by measuring uptake of 68Ga-DOTANOC with PET/CT in patients with newly diagnosed non-Hodgkin's and Hodgkin's lymphoma. The imaging findings will be compared to immunohistochemically determined ssr-subtypes 2,3 and 5 obtained from pre-treatment fresh tumor samples and 18F-FDG PET/CT which is part of standard diagnostic evaluation. Furthermore, whole-body MRI with DWI will be performed before, during and after chemotherapy to define the most sensitive and specific imaging method appropriate for routine diagnosis and follow-up. This study has potential implications for future response monitoring and follow-up imaging techniques in patients with malignant lymphoma and provides additional biologic characterization which may be useful for novel therapeutic approaches such as PRRT.

DETAILED DESCRIPTION:
Lymphomas are malignant tumours of the immune system. Lymphomas are classified as Hodgkin's or non-Hodgkin's lymphomas with several subtypes. In Finland the amount of newly diagnosed Hodgkin's lymphomas is 120-150 new cases per year and it accounts for 12 % of all lymphomas. Non-Hodgkin's lymphoma is the sixth most common cancer in men and the eight most common cancer in women in Finland. There are approximately 1200 new cases per year and the incidence has been increasing during the last decade. (1, 2)

Etiology of lymphomas is mostly unknown but many risk factors have been identified. Diagnostics and classification to different subgroups is based on clinical, pathological, molecular, and radiological studies. Some of lymphoma's subtypes can be cured with current treatment methods, however, many of them remain still incurable. (1) Clearly, more accurate diagnostic tools with subsequent targeted therapies against lymphomas are needed.

Somatostatin receptors (SSTs) are expressed by a wide variety of different tumour cell types, including malignant lymphomas. (8, 9, 10, 11) Somatostatin receptor imaging by octreotide scintigraphy has showed a sensitivity of 95-100 % in Hodgkin's lymphoma and 80 % in non-Hodgkin's lymphoma. However, somatostatin receptor scintigraphy does not appear to have a significant role in diagnostic process because of the relatively low uptake of the used somatostatin analogue (octreotide) and limited sensitivity of the single photon emission computed tomography (SPECT) acquisition to detect and localise small involved nodes. (11, 25) Hence, somatostatin receptor imaging has been further developed with the advent of hybrid SPECT and positron emission tomography (PET) and computed tomography (CT) scanners. Several other radioligands have been studied to improve the binding affinity (15). This has also offered a new target for tumor cell-specific therapy using different somatostatin analogs labelled with therapeutic radionuclides such as 90Y-DOTATOC, a somatostatin receptor subtype 2 (SST2) -specific ligand. Clinical studies of peptide receptor radionuclide therapy (PRRT) have extensively focused on neuroendocrine tumors as a palliative treatment modality (12, 13, 14). Another new candidate for SST based imaging and treatment is 68Ga-DOTANOC, a high-affinity ligand of somatostatin receptor subtypes 2, 3 and 5 (SST2, SST3, SST5) (16). Neuroendocrine tumors are known to express SST2 and they show high uptake of radiolabeled somatostatin analogs on PET. However, lymphomas may mimick NETs on DOTANOC PET/CT as was shown in a recent case report (17). Therefore, further studies on SST2 status and DOTANOC uptake are in order to establish the role of peptide based imaging in diagnosis and possible PRRT in lymphomas.

The aim of the study is to determine tumor uptake of 68Ga-DOTANOC in patients with non-Hodgkin's and Hodgkin's lymphoma to characterize the SST2, SST3 and SST5 receptor status of the tumour in vivo with 68Ga-DOTANOC PET/CT. In addition, immunohistochemical analysis of SST2, SST3 and SST5 subtype status will be made of the tumor specimens obtained in routine diagnostic biopsy resection. Furthermore, PET findings will be correlated with advanced MRI techniques, such as diffusion weighted imaging (DWI) in an attempt to find methods which limit radiation exposure especially in young patients. Hence, PET/CT will be performed with 68Ga-DOTANOC and 18F-FDG and compared with whole-body MRI (including DWI) to define the most sensitive and specific imaging method appropriate for routine diagnosis and follow-up of patients with lymphoma.

To the investigators knowledge, no prospective studies comparing octreodite analogue based PET/CT imaging with standard diagnostic procedures have been published until now. PET/CT offers a clear advantage over scintigraphy in terms of sensitivity and resolution which should be helpful in determining the SST status of various histologic forms of lymphomas The investigators hypothesize that a positive 68Ga-DOTANOC PET/CT scan correlates with the overexpression of all or some SST subtypes in lymphomas, which is possibly linked to a more indolent behavior of the disease. Furthermore, it is hypothesized that 68Ga-DOTANOC PET/CT imaging provides a valid method to select patients with lymphoma for radionuclide therapy with 177Lu-DOTATATE. Third, differential diagnosis with NETs may also improve after receiving information on SST status in lymphomas. Thus findings in this study may be useful not only for biologic characterization but also for diagnosis and management of these heterogenous diseases originating in the lymphatic system

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old
* Language spoken: Finnish or Swedish
* Patients with diagnosed untreated non-Hodgkin's or Hodgkin's lymphoma with measurable disease (the diagnosis is based on radiological, histological and clinical grounds)
* Before treatment CT and FDG-PET performed
* Mental status: Patients must be able to understand the meaning of the study
* The patient signs the appropriate Ethical Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Any medical or psychiatric condition that compromises the subject's ability to participate in the study
* Any other significant disease including liver or renal disease
* Pregnant or lactating women
* Contraindications for MR imaging

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Knuuti, M.D., Ph.D., Study Chair — Turku PET Centre
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] Ferlay J, Autier P, Boniol M, Heanue M, Colombet M, Boyle P. Estimates of the cancer incidence and mortality in Europe in 2006. Ann Oncol. 2007 Mar;18(3):581-92. doi: 10.1093/annonc/mdl498. Epub 2007 Feb 7. PMID 17287242
- [Background] Gallamini A, Borra A. Role of PET in lymphoma. Curr Treat Options Oncol. 2014 Jun;15(2):248-61. doi: 10.1007/s11864-014-0278-4. PMID 24619427
- [Background] Mayerhoefer ME, Karanikas G, Kletter K, Prosch H, Kiesewetter B, Skrabs C, Porpaczy E, Weber M, Pinker-Domenig K, Berzaczy D, Hoffmann M, Sillaber C, Jaeger U, Mullauer L, Simonitsch-Klupp I, Dolak W, Gaiger A, Ubl P, Lukas J, Raderer M. Evaluation of diffusion-weighted MRI for pretherapeutic assessment and staging of lymphoma: results of a prospective study in 140 patients. Clin Cancer Res. 2014 Jun 1;20(11):2984-93. doi: 10.1158/1078-0432.CCR-13-3355. Epub 2014 Apr 2. PMID 24696320
- [Background] Reubi JC, Waser B, van Hagen M, Lamberts SW, Krenning EP, Gebbers JO, Laissue JA. In vitro and in vivo detection of somatostatin receptors in human malignant lymphomas. Int J Cancer. 1992 Apr 1;50(6):895-900. doi: 10.1002/ijc.2910500613. PMID 1348240
- [Background] Lugtenburg PJ, Krenning EP, Valkema R, Oei HY, Lamberts SW, Eijkemans MJ, van Putten WL, Lowenberg B. Somatostatin receptor scintigraphy useful in stage I-II Hodgkin's disease: more extended disease identified. Br J Haematol. 2001 Mar;112(4):936-44. doi: 10.1046/j.1365-2141.2001.02583.x. PMID 11298588
- [Background] Ferone D, Hofland LJ, Colao A, Lamberts SW, van Hagen PM. Neuroendocrine aspects of immunolymphoproliferative diseases. Ann Oncol. 2001;12 Suppl 2:S125-30. doi: 10.1093/annonc/12.suppl_2.s125. PMID 11762338
- [Background] Ferone D, Semino C, Boschetti M, Cascini GL, Minuto F, Lastoria S. Initial staging of lymphoma with octreotide and other receptor imaging agents. Semin Nucl Med. 2005 Jul;35(3):176-85. doi: 10.1053/j.semnuclmed.2005.03.001. PMID 16098291
- [Background] Kwekkeboom DJ, Mueller-Brand J, Paganelli G, Anthony LB, Pauwels S, Kvols LK, O'dorisio TM, Valkema R, Bodei L, Chinol M, Maecke HR, Krenning EP. Overview of results of peptide receptor radionuclide therapy with 3 radiolabeled somatostatin analogs. J Nucl Med. 2005 Jan;46 Suppl 1:62S-6S. PMID 15653653
- [Background] Reubi JC, Schar JC, Waser B, Wenger S, Heppeler A, Schmitt JS, Macke HR. Affinity profiles for human somatostatin receptor subtypes SST1-SST5 of somatostatin radiotracers selected for scintigraphic and radiotherapeutic use. Eur J Nucl Med. 2000 Mar;27(3):273-82. doi: 10.1007/s002590050034. PMID 10774879
- [Background] Wild D, Schmitt JS, Ginj M, Macke HR, Bernard BF, Krenning E, De Jong M, Wenger S, Reubi JC. DOTA-NOC, a high-affinity ligand of somatostatin receptor subtypes 2, 3 and 5 for labelling with various radiometals. Eur J Nucl Med Mol Imaging. 2003 Oct;30(10):1338-47. doi: 10.1007/s00259-003-1255-5. Epub 2003 Aug 21. PMID 12937948
- [Background] Jain S, Sharma P, Dhull VS, Bal C, Kumar R. Lymphoma as a second malignancy in a patient with neuroendocrine tumor: mimicking dedifferentiation on dual-tracer PET/CT with 68Ga-DOTANOC and 18F-FDG. Clin Nucl Med. 2014 Apr;39(4):358-9. doi: 10.1097/RLU.0b013e31828e98c5. PMID 24217543

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lymphoma
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with lymphoma
Groups:
- Study Patients: Patiens with lymphoma
Arm/Group | Study Patients
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] — One 82-year old patient was included which exceeded the upper age limit specified in the inclusion criteria because of a protocol violation
  years | 66 [40 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: 68Ga-DOTANOC Uptake in Lymphomas With PET/CT
Description: Uptake of 68Ga-DOTANOC in lymphoma expressed as SUVmax
Time Frame: Within 30 days prior to start of chemotherapy
Population: Lesion with highest radioactivity
Measure: Median (Full Range); unit: Standardized Uptake Value
Units Other Than Participants: Lymphomatous lesion
Groups:
- Lymphoma: Uptake of 68Ga-DOTANOC
Arm/Group | Lymphoma
Number analyzed (Participants) | 21
Number analyzed (Lymphomatous lesion) | 21
Standardized Uptake Value | 3.1 [1.9 to 9.8]

ADVERSE EVENTS:
Arm/Group | Lymphoma
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No